CLINICAL TRIAL: NCT00275587
Title: Development of Critical Pathway Care for Hospitalized Patients Using Principles of Patient-Centered Quality Care, Evidence-Based Medicine, and High Reliability Organizational Structure
Brief Title: Development of a Hospital Service That Uses Critical Pathway (Protocolized) Care Plans to Provide High-Quality, High-Reliability, Evidence-Based Medical Care
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: A. Scott Keller, Mayo Clinic
Other Study IDs: 164-05
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Critical Pathways

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Our broad, long-term objective is to create a new non-resident (non-teaching) hospital service that uses patient-centered critical pathway care plans for treating patients in St. Marys Hospital. This innovative service, the Hospital Medicine (HOME) Team, will integrate three timely, high-priority concepts in healthcare: patient-centered quality care, evidence-based medicine, and principles that define high reliability organizations. The target populations for the new model of service are patients hospitalized with pre-defined admission diagnoses who are expected to require only a brief, focused hospital stay of four days or less. Specifically, we will 1) Design the prototypical approach to be used for developing all critical pathway care plans by integrating patient-centered quality care, evidence-based medicine, and principles that define high reliability organizations, 2) Systematically design the critical pathway care plans for two pre-defined admission diagnoses (community-acquired pneumonia and non-surgical low-back pain), and 3) Compare outcomes of this new service against respective historical patient cohorts for patients admitted with community-acquired pneumonia and non-surgical low-back pain. We anticipate that the prototypic methodology used to develop this patient-centered service will be replicated for other new hospital-service models. To our knowledge, there are currently no existing hospital services in the U.S. that have intentionally integrated principles of high reliability organizations into evidence-based critical pathways founded on patient-centered principles of uncompromising quality.

ELIGIBILITY:
1. Hospitalized patient with one of six medical diagnoses: community-acquired pneumonia, deep venous thrombosis or pulmonary embolism, cellulitis, alcohol withdrawal, pyelonephritis, low back pain.
2. Ability and agreement to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at St. Marys Hospital in Rochester, MN with with one of six medical diagnoses: community-acquired pneumonia, deep venous thrombosis or pulmonary embolism, cellulitis, alcohol withdrawal, pyelonephritis, low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Scott Keller, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States